CLINICAL TRIAL: NCT00163449
Title: BALLOON: Efficacy and Safety - Study by ALTANA on Ciclesonide in Pre-school Asthma Patients
Brief Title: Efficacy and Safety of Ciclesonide in Preschool Children With Asthma (2 to 6 Years) (BY9010/M1-207)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BY9010/M1-207
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Child; Pediatric
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 1 (Active Comparator): Ciclesonide 40 µg
  Interventions: Drug: Ciclesonide
- 2 (Active Comparator): Ciclesonide 80 µg
  Interventions: Drug: Ciclesonide
- 3 (Active Comparator): Ciclesonide 160 µg
  Interventions: Drug: Ciclesonide
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — Efficacy and Safety of Ciclesonide
  Arms: 1; 2; 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
The aim of the present study is to compare the efficacy of inhaled ciclesonide in pre-school children. Ciclesonide will be inhaled once daily, using one of three dose levels and tested versus placebo. The study duration consists of a baseline period (2 to 4 weeks) and a treatment period (24 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent by the parents or legal guardians of the patient
* Outpatients
* Good health with the exception of asthma
* Documented diagnosis of asthma for more than 6 months
* Use of rescue medication only or pretreatment with a controller drug

Main Exclusion Criteria:

* Concomitant severe diseases
* Diseases contraindicated for the use of inhaled steroids
* Other relevant lung diseases causing impairment in pulmonary function
* Recurrent, episodic wheezing only
* History of life-threatening asthma
* History of any mechanical ventilation
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation
* Premature birth (< 32 weeks gestation)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
time to first moderate or severe asthma exacerbation. | 24 weeks

SECONDARY OUTCOMES:
rate of patients with moderate or severe asthma exacerbation | 24 weeks
rate of patients with moderate asthma exacerbation | 24 weeks
rate of patients with severe asthma exacerbation | 24 weeks
time to first moderate asthma exacerbation | 24 weeks
time to first severe asthma exacerbation | 24 weeks
asthma symptom score from diary | 24 weeks
use of rescue medication | 24 weeks
patient perceived asthma control | 24 weeks
quality of life data (PACQLQ) | 24 weeks
morning and evening PEF from diary | 24 weeks
pulmonary function variables measured at the investigational sites | 24 weeks
adverse events | 24 weeks
physical examination | 24 weeks
vital signs | 24 weeks
laboratory work-up | 24 weeks
serum cortisol | 24 weeks
urine cortisol variables | 24 weeks
body growth determined by stadiometry. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (82):
- Brazil (14):
  - Altana Pharma/Nycomed, Campinas - SP
  - Altana Pharma/Nycomed, Curitiba-PR
  - Altana Pharma/Nycomed, Paraná
  - Altana Pharma/Nycomed, Pinheiros Sao Paulo - SP
  - Altana Pharma/Nycomed, Porto Alegre-RS
  - Altana Pharma/Nycomed, Recife-PE
  - Altana Pharma/Nycomed, Rio de Janeiro-RJ
  - Altana Pharma/Nycomed, Rio Grande
  - Altana Pharma/Nycomed, Salvador - Bahia
  - Altana Pharma/Nycomed, Santo André-SP
  - Altana Pharma/Nycomed, Sao Paulo - SP
  - Altana Pharma/Nycomed, Sao Paulo-SP
  - Altana Pharma/Nycomed, São Paulo
  - Altana Pharma/Nycomed, São Paulo-SP
- Germany (11):
  - Altana Pharma/Nycomed, Berlin
  - Altana Pharma/Nycomed, Cologne
  - Altana Pharma/Nycomed, Dresden
  - Altana Pharma/Nycomed, Düsseldorf
  - Altana Pharma/Nycomed, Frankfurt
  - Altana Pharma/Nycomed, Heidelberg
  - Altana Pharma/Nycomed, Mannheim
  - Altana Pharma/Nycomed, München
  - Altana Pharma/Nycomed, Rosenheim
  - Altana Pharma/Nycomed, Wesel
  - Altana Pharma/Nycomed, Wiefelstede
- Hungary (14):
  - Altana Pharma/Nycomed, Baja
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Debrecen
  - Altana Pharma/Nycomed, Jászberény
  - Altana Pharma/Nycomed, Kaposvár
  - Altana Pharma/Nycomed, Kiskunhalas
  - Altana Pharma/Nycomed, Miskolc
  - Altana Pharma/Nycomed, Mosdós
  - Altana Pharma/Nycomed, Mosonmagyaróvár
  - Altana Pharma/Nycomed, Nyíregyháza
  - Altana Pharma/Nycomed, Pécs
  - Altana Pharma/Nycomed, Szeged
  - Altana Pharma/Nycomed, Szekszárd
  - Altana Pharma/Nycomed, Törökbálint
- India (10):
  - Altana Pharma/Nycomed, Chandanwadi, Thane
  - Altana Pharma/Nycomed, Chennai
  - Altana Pharma/Nycomed, Coimbatore
  - Altana Pharma/Nycomed, Coimbatore, Tamilnadu
  - Altana Pharma/Nycomed, Kalaburagi
  - Altana Pharma/Nycomed, Mumbai
  - Altana Pharma/Nycomed, Mumbai, Dadar (E)
  - Altana Pharma/Nycomed, Nagpur
  - Altana Pharma/Nycomed, Noida
  - Altana Pharma/Nycomed, Pune
- Netherlands (6):
  - Altana Pharma/Nycomed, Eindhoven
  - Altana Pharma/Nycomed, Enschede
  - Altana Pharma/Nycomed, Hoofddorp
  - Altana Pharma/Nycomed, Leeuwarden
  - Altana Pharma/Nycomed, Nijmegen
  - Altana Pharma/Nycomed, Zwolle
- Poland (5):
  - Altana Pharma/Nycomed, Karpacz
  - Altana Pharma/Nycomed, Lublin
  - Altana Pharma/Nycomed, Opole
  - Altana Pharma/Nycomed, Poznan
  - Altana Pharma/Nycomed, Zawadzkie
- South Africa (11):
  - Altana Pharma/Nycomed, Bellville - Cape Town -
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, Durban
  - Altana Pharma/Nycomed, Morningside, Sandton
  - Altana Pharma/Nycomed, Mowbray, Cape Town
  - Altana Pharma/Nycomed, New Redruth, Alberton
  - Altana Pharma/Nycomed, Overport, Durban
  - Altana Pharma/Nycomed, Panorama / RSA-Cape Town
  - Altana Pharma/Nycomed, Pietermaritzburg
  - Altana Pharma/Nycomed, Westville
  - Altana Pharma/Nycomed, Wynberg
- Spain (8):
  - Altana Pharma/Nycomed, Barcelona
  - Altana Pharma/Nycomed, El Palmar (Murcia)
  - Altana Pharma/Nycomed, Elche - Alicante
  - Altana Pharma/Nycomed, Leganes (Madrid)
  - Altana Pharma/Nycomed, Madrid
  - Altana Pharma/Nycomed, Sabadell
  - Altana Pharma/Nycomed, Seville
  - Altana Pharma/Nycomed, Valencia
- Switzerland (3):
  - Altana Pharma/Nycomed, Lausanne
  - Altana Pharma/Nycomed, Trimbach
  - Altana Pharma/Nycomed, Zurich

REFERENCES:
- [Derived] Brand PL, Luz Garcia-Garcia M, Morison A, Vermeulen JH, Weber HC. Ciclesonide in wheezy preschool children with a positive asthma predictive index or atopy. Respir Med. 2011 Nov;105(11):1588-95. doi: 10.1016/j.rmed.2011.07.017. Epub 2011 Aug 11. PMID 21839625
- See also: BY9010-M1-207-DEU RDS-2008-03-20.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4527&filename=BY9010-M1-207-DEU%20RDS-2008-03-20.pdf